CLINICAL TRIAL: NCT02727478
Title: Highly Challenging Balance Training for People With Parkinson's Disease (the BETA-PD Study): Non-randomized Hybrid Effectiveness-implementation Trial
Brief Title: Effectiveness and Implementation of the HiBalance Program in Clinical Practice
Acronym: BETA-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Erika Franzén, Associate Professor, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/210-31/2
Record Dates: First submitted 2016-03-22; First posted 2016-04-04 (Estimated); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease
Keywords: Balance; Rehabilitation; Exercise; basal ganglia; Gait; Training; physical activity
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balance training group (Experimental): 1 hour group balance training twice weekly for 10 weeks, as well as perform a home exercise program.
  Interventions: Other: HiBalance training program
- Control group (No Intervention): Subjects in this group will receive no intervention and will be advised to continue their normal level of exercise throughout the intervention period.

INTERVENTIONS:
Other: HiBalance training program — The program consists of physiotherapist led highly challenging balance exercises, which are adapted and progressed on both a group and individual basis throughout the training period.
  Arms: Balance training group

SUMMARY:
This effectiveness-implementation study is a part of the larger study BETA-PD (Balance, Elderly, Training and Activity in Parkinson's Disease), which has the long-term goal to reduce the risk of falling in people with Parkinson's disease (PD) by improving balance, gait and physical activity level. The main hypothesis is that highly challenging balance training will lead to greater gait and balance ability, increased levels of physical activity and an improved health related quality of life. The main aims of the study are to evaluate the effectiveness of the HiBalance program in real-life clinical settings, while exploring facilitators and barriers for program implementation on a wider scale.

DETAILED DESCRIPTION:
The clinical features of PD include progressive postural instability, hypokinesia, tremor and rigidity. It is therefore common that people with PD experience reduced balance and gait function, symptoms which can have far-reaching negative effects on their health and quality of life. Injurious falls and fear of falling are especially prevalent among those with PD, a factor which may partly explain why this group are less physically active than older people of a similar age without the diagnosis. Balance and gait training, on the other hand, have been shown effective in PD and also appear to have potential neuro-protective properties. Research in the area of balance training in PD disease however is sparse and previous interventions have been criticized for applying training stimuli which lacked intensity and challenge.

The HiBalance program is based on scientifically well-established principles of exercise training and postural control as well as current research on training in PD. The program was developed to affect symptom-specific balance impairments in PD by targeting four main subsystems underlying balance control (stability limits, anticipatory postural adjustments, sensory integration and motor agility). The intervention consists of a 10-week progressive balance training program in group format (5-7 participants). Each training session is conducted by a minimum of 2 physiotherapist trainers, during twice weekly 1-hour sessions (20 hours in total). Additionally, a home-exercise program is carried out by the participants once a week during the trial period. The difficulty level of the group-based training is increased in three consecutive blocks. To ensure highly challenging exercises, each task is individually adjusted by altering the area of base of support, increasing movement speed/amplitude and/or restricting vision and varying the grade of multitasking. The program has previously been proven feasible [Conradsson, 2012] and effective [Conradsson, 2015] in improving balance and gait impairments in a randomized controlled hospital setting. In addition, favorable transfer effects were seen in relation to physical activity levels and the performance of activities of everyday life.

For research interventions to be adopted in real-life clinical settings however a level of adaptation is required. Best practice then involves evaluating the effectiveness of efficacious programs in clinical settings, in order to verify whether or not the adaptation has attenuated the effective core elements of the program itself.

The current study combines a clinical effectiveness trial together with implementation research. Use of a type-1 hybrid design will allow the effects of the HiBalance program in clinical settings to be tested while simultaneously gathering information on barriers and facilitators to the implementation process [Curran, 2012]. Use of the hybrid design also allows for constant monitoring of the process by which the intervention is applied, and therefore allow problems in early application to be identified and quickly altered so as to ensure better outcomes. A participatory approach will be adhered to whereby 'users' of the program (physiotherapist trainers) will be actively involved in all stages of the program adaptation, process and outcome evaluation. This approach is recommended in order to increase the relevance, acceptability and successful implementation of the program. The Consolidated Framework for Implementation Research (CFIR) will be used in the current study to guide the investigation of potential barriers to and facilitators of the implementation process [Damschroder, 2009 ].

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed idiopathic Parkinson's Disease
* Measured balance impairment (according to the mini-BESTest)
* Hoehn and Yahr stages 2-3
* Independent ambulator indoors without a walking aid

Exclusion Criteria:

* Cognitive impairment which hinders participation in group training
* The presence of comorbidities which hinder safe participation in group training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erika Franzén, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska institutet, Stockholm, Södermanland County, Sweden

REFERENCES:
- [Background] Conradsson D, Lofgren N, Stahle A, Hagstromer M, Franzen E. A novel conceptual framework for balance training in Parkinson's disease-study protocol for a randomised controlled trial. BMC Neurol. 2012 Sep 27;12:111. doi: 10.1186/1471-2377-12-111. PMID 23017069
- [Background] Conradsson D, Lofgren N, Nero H, Hagstromer M, Stahle A, Lokk J, Franzen E. The Effects of Highly Challenging Balance Training in Elderly With Parkinson's Disease: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2015 Oct;29(9):827-36. doi: 10.1177/1545968314567150. Epub 2015 Jan 21. PMID 25608520
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Result] Leavy B, Joseph C, Lofgren N, Johansson H, Hagstromer M, Franzen E. Outcome Evaluation of Highly Challenging Balance Training for People With Parkinson Disease: A Multicenter Effectiveness-Implementation Study. J Neurol Phys Ther. 2020 Jan;44(1):15-22. doi: 10.1097/NPT.0000000000000298. PMID 31834166
- [Derived] Leavy B, Joseph C, Kwak L, Franzen E. Implementation of highly challenging balance training for Parkinson's disease in clinical practice: a process evaluation. BMC Geriatr. 2021 Feb 1;21(1):96. doi: 10.1186/s12877-021-02031-1. PMID 33526031
- [Derived] Leavy B, Kwak L, Hagstromer M, Franzen E. Evaluation and implementation of highly challenging balance training in clinical practice for people with Parkinson's disease: protocol for the HiBalance effectiveness-implementation trial. BMC Neurol. 2017 Feb 7;17(1):27. doi: 10.1186/s12883-017-0809-2. PMID 28173775

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Balance Training Group | Control Group
Started | 61 | 56
Completed | 53 | 46
Not Completed | 8 | 10
Not completed — Withdrawal by Subject | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Balance Training Group | Control Group | Total
Number analyzed (Participants) | 61 | 56 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (8.5) | 70 (6.5) | 70. (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 22 | 55
  Male | 28 | 34 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 61 | 56 | 117

OUTCOME MEASURES:

1. Primary Outcome: Change in Mini-BESTest Score From Baseline at 1 Week Post Intervention.
Description: Mini-Balance Evaluation Systems Test a rating scale for dynamic balance incorporating 14 different balance and gait items that were assessed by a physical therapist on a scale from 0-2. Maximum points 28.
  0-28 points with higher scores indicating better balance control The mini-BESTest is an assessment of balance performance and will be performed by the physiotherapists in the respective clinics.
Time Frame: Change in Mini-BESTest score from baseline at 1 week post intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Balance Training Group | Control Group
Number analyzed (Participants) | 61 | 56
score on a scale | 2.0 (2.0) | -0.2 (2.4)
Statistical Analysis 1: Comparison: Balance Training Group vs Control Group; Test type: Superiority; p < 0.001, ANOVA

2. Secondary Outcome: Change in 10-meter Walking Test Score From Baseline at 1 Week Post Intervention.
Description: The 10-meter walking test assesses gait performance was performed by the physiotherapists in the respective clinics.
  Gait speed was measured as m/sec during 10 meters
Time Frame: From baseline at 1 week post intervention.
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Balance Training Group | Control Group
Number analyzed (Participants) | 60 | 56
m/sec | 0.2 (0.41) | -0.04 (0.14)
Statistical Analysis 1: Comparison: Balance Training Group vs Control Group; Test type: Superiority; p = 0.001, ANOVA

3. Secondary Outcome: Change in Timed Up and Go (TUG) Test From Baseline at 1 Week Post Intervention.
Description: The TUG test assesses functional mobility and will be performed by the physiotherapists in the respective clinics. TUG test measures performance of a sequential locomotor task (rising from a chair, walking 3 m, turning and walking back to the chair). Timed Up and Go (TUG) test is measured in seconds it takes to perform the task.
Time Frame: From baseline at 1 week post intervention.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Balance Training Group | Control Group
Number analyzed (Participants) | 61 | 56
seconds | -0.4 [-1.13 to 0.5] | 0 [-1.6 to 1.2]
Statistical Analysis 1: Comparison: Balance Training Group vs Control Group; Test type: Other; p = 0.254, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in EQ-5D Score From Baseline at 1week Post Intervention.
Description: The EQ-5D is a 2-paged form assessing health-related quality of life and will be filled in by participants.
  European Quality of Life- 5 dimensions (EQ-5D), The visual analogue scale (VAS) indicates the general health status ranging from 0-100 with 100 indicating the best health status
Time Frame: From baseline at 1week post intervention.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Balance Training Group | Control Group
Number analyzed (Participants) | 59 | 48
units on a scale | 5.5 [-5 to 15] | 0 [-10 to 5]
Statistical Analysis 1: Comparison: Balance Training Group vs Control Group; Test type: Superiority; p = 0.065, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Activities-specific Balance Confidence (ABC) Scale
Description: The ABC scale assesses self-reported balance confidence and will be filled in by study participants.
  It consists of 16 items that are rated from from 0-100% where 0% indicates no confidence and 100% complete confidence.
  The overall score is calculated by adding the item scores and dividing the total by 16 (i.e. the number of items). This total score ranges from 0% to 100%.
Time Frame: From baseline at 1 week post intervention.
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Balance Training Group | Control Group
Number analyzed (Participants) | 60 | 47
units on a scale | 68 (16.9) | 70 (18.2)
Statistical Analysis 1: Comparison: Balance Training Group vs Control Group; Test type: Superiority; p = 0.301, ANOVA

6. Secondary Outcome: Change in Physical Activity Level From Baseline 1 Week Post Intervention.
Description: Participants will wear accelerometers for a 7-day period directly before and after the intervention.
  Physical activity level (steps per day)
Time Frame: from baseline to 1 week post intervention
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Balance Training Group | Control Group
Number analyzed (Participants) | 53 | 48
steps per day | -288 (1428) | -390 (2016)
Statistical Analysis 1: Comparison: Balance Training Group vs Control Group; Test type: Superiority; p = 0.792, ANOVA

7. Secondary Outcome: Change in Dual Task Interference During the Timed Up and Go (TUG) Test From Baseline at 1 Week Post Intervention.
Description: The TUG test assesses functional mobility and will be performed by the physiotherapists in the respective clinics.
  TUG test measures performance of a sequential locomotor task (rising from a chair, walking 3 m, turning and walking back to the chair).The TUG COG test involves performance of the TUG test while sequentially subtracting the number 3 from a start number. The time difference between the TUG and the TUG COG reflects dual-task interference during functional mobility and is calculated be expressed as a percentage: (TUG COG - TUG)/TUG.
Time Frame: From baseline at 1 week post intervention.
Measure: Median (Inter-Quartile Range); unit: percentage of interference
Arm/Group | Balance Training Group | Control Group
Number analyzed (Participants) | 53 | 55
percentage of interference | -1.22 [-6.2 to 0.66] | 1.05 [-3.07 to 3.51]
Statistical Analysis 1: Comparison: Balance Training Group vs Control Group; Test type: Other; p = 0.039, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: Adverse events collected through observation during the training sessions. All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed for the Control Group.
Arm/Group | Balance Training Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/0
Other Adverse Events (participants affected / at risk) | 12/61 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balance Training Group (N=61) | Control Group (N=0)
Falls (Injury, poisoning and procedural complications) | 12 (12) | 0 (0) — 12 non-injurious falls occurred during the training sessions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT02727478/Prot_SAP_000.pdf